CLINICAL TRIAL: NCT02861794
Title: Evaluation of Early Migration of Medially Stabilized Arthroplasty as a Predictor of Long Time Survivorship (Implant Design Study)
Brief Title: Stability of Contemporary Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Helse More and Romsdal Trust (Unknown); Medacta International SA (Industry)
Responsible Party: Principal Investigator, Stephan M Rohrl, Ass. professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 424444-1
Record Dates: First submitted 2016-04-28; First posted 2016-08-10 (Estimated); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
Keywords: Total Knee Arthroplasty (TKA); Total Knee Replacement (TKR); Kinematics; RSA; Knee arthroplasty; Implant stability; Migration; Wear; Medial pivot
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective interventional single group cohort study of a cemented medial pivot knee implant, using the diagnostic method of RSA.
Masking Description: Non-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GMK Sphere (Other): Patients receive a GMK Sphere Total Knee Replacement.
  Interventions: Procedure: Medacta International, GMK Sphere medially stabilized knee

INTERVENTIONS:
Procedure: Medacta International, GMK Sphere medially stabilized knee — Total Knee Replacement

SUMMARY:
Total joint replacement is an efficacious treatment for osteoarthritis of hips and knees. Both total knee replacement (TKR) and total hip replacements (THR) have excellent implant survivorship. However, patient satisfaction is lower in TKR than THR. A possible cause of the discrepancy is the unnatural knee kinematics after TKR. Various implants designs have been developed to solve the problem. However, most of their designs are based on experimental data and little has been studied about their actual performance in vivo. In this study, the investigators will analyze the in vivo stability of the Global Medacta Knee Sphere (GMK Sphere) implant. Migration of the implants will be monitored with a high precision measuring method called Radiostereometric Analysis (RSA). The investigators assume the investigators study will contribute the development of more satisfying knee implants.

DETAILED DESCRIPTION:
Worldwide the number of patients requiring treatment for osteoarthritis is increasing due to increasing obesity, an ageing population and a high demanding younger population. Learmonth describes hip arthroplasty as the "operation of the century" because patients are highly satisfied with pain relief and function after the procedure. Knee arthroplasties have in recent years also shown promising results and have surpassed hip arthroplasty in frequency in western countries. However, patient satisfaction is not as high. Reported problems are insufficient function and persistent pain. On the other hand, knee arthroplasties are increasingly implanted in younger and more active patients who require high function and quality of life. Improvement of knee implants is an urgent issue in the field of orthopaedic research.

Knee Kinematics and implant designs

A possible cause of lower function of replaced knees is the unnatural postoperative knee kinematics. Kinematics of replaced knees is closely related to their function. Studies show that replaced knees with excellent flexion angles have kinematic similarities to normal knees and malalignments of implants can cause postoperative pain.

Compared to hip joints which are simple ball-and socket joints, the kinematics of knee joints is more complex. The kinematics are a combination of a rolling and gliding motion of the femoral condyles and rotation of the tibia. Based on the kinematics of the normal knee joint, various attempts have been made on the design of knee implants to reconstruct normal kinematics after replacement surgery. All of these implants have satisfying survivorship, but unicondylar arthroplasty which retains both cruciate ligaments has the best clinical results with survivorship at 15 years 93%. In total knee replacement (TKR) the Anterior Cruciate Ligament (ACL) and possibly the Posterior Cruciate Ligament (PCL) are sacrified. When sacrificing the one or both of the cruciate ligaments, natural knee kinematics are affected. The function of the cruciate ligaments can be mimicked by different designs of the tibial insert.

The most used knee implant in Norway, the NexGen Cruciate-retaining (CR) implant design, does not retain the ACL and does not mimic natural knee kinematics. The tibial insert of the medial pivot implant design (GMK Sphere) has a constrained medial ball in socket joint and at the same time allows lateral anterioposterior movement. This new design was developed by a group of dedicated researchers. The design intention is to resemble the function of the cruciate ligaments and at the same time allow for lateral anterioposterior movement (rollback).

Small alterations in implant design can influence the survival of implants. The final design of the GMK Sphere was introduced in 2012. New implants should be monitored and assessed in small, controlled trials with high precision measuring methods.

Analytical Method

RSA has been used in orthopedic research fields since 1970s. The original application of this method was for the evaluation of implant migration (i.e. fixation) and polyethylene wear of artificial joints using static X-ray pictures. Clinically relevant association between early migration of tibial implants detected by RSA and late revision for loosening has been reported. Also, attempts to measure in vivo polyethylene wear have been reported using RSA.

Purpose of this study

The aim of this study is to analyse the in vivo performance (e.g. stability) of a medially stabilized knee arthroplasty implant (Medacta International, GMK Sphere) using static RSA method over a period of 5 years. 2-year results have already been analysed and are inconclusive in regards to migration as the implant is apparently stable, but shows greater than anticipated movement. Mid-term follow-up (5-year) is therefore essential to evaluate migration of this implant. We therefore wish to obtain 5-year follow-ups of these patients.

Additionally, the investigators will analyse the wear in the ball and socket (medial) side of the tibiofemoral articulation.

30 patients will go through stability and wear testing with static RSA.

This study will contribute to the safety for patients with this new implant by providing basic knowledge of this knee arthroplasty and promoting further development of knee implant designs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with knee osteoarthritis

Exclusion Criteria:

* Preoperative severe deformity (Femoro-tibial angle < 175°or > 190°measured on a full-length leg image at weight bearing)
* Preoperative flexion contracture more than 15°
* Preoperative limited range of motion under anesthetics (less than 110°)
* Less than 50 or more than 75 years of age at the time of surgery
* Use of walking aids because of other musculoskeletal and neuromuscular problems
* Preoperative diagnosis other than osteoarthritis and avascular necrosis (e.g. rheumatoid arthritis, tumors)
* Revision arthroplasty
* Obesity with BMI >35
* Impaired collateral ligaments
* Malposition of femoral and tibial implants (Internally rotated or more than 10° externally rotated implants will be excluded. The rotation of femoral implant is measured on postoperative CT images in reference to surgical epicondylar line. The rotation of tibial implant is determined according to Berger's measurement)
* Postoperative revision surgery due to deep wound infection

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stability of the GMK Sphere prosthesis measured by Radiostereometric Analysis (RSA) | 5 years
  Stability of the implant is measured in mm after 5 years (Maximum Total Point Motion in mm, MTPM)

SECONDARY OUTCOMES:
Knee Society Score (KSS) | 5 years
  Patient reported outcome measures
Forgotten Joint Score 12 (FJS-12) | 5 years
  Patient reported outcome measures
Knee injury and Osteoarthritis Outcome Score (KOOS) | 5 years
  Patient reported outcome measures
Range of motion (ROM) | 5 years
  Clinical measurement using goniometer
Hip-knee-ankle angle (HKA-angle) | 5 years
  The axis of the lower extremity after knee arthroplasty
CT-rotation of implants | 5 years
  Evaluation of tibia implant rotation using Berger's method
Stability of the GMK Sphere prosthesis | 5 years
  Stability of the implant is measured in mm and degrees after 5 years using RSA (translation and rotasjon for x, y and z)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Maximillian Røhrl, MD, PhD, Study Director — Center for Implant and Radiostereometric Research Oslo (CIRRO); Frank-David Oehrn, MD, Principal Investigator — Kristiansund Hospital, Helse More and Romsdal Trust; Lars Harald William Engseth, MD, PhD, Principal Investigator — Center for Implant and Radiostereometric Research Oslo (CIRRO)
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Kurtz SM, Lau E, Ong K, Zhao K, Kelly M, Bozic KJ. Future young patient demand for primary and revision joint replacement: national projections from 2010 to 2030. Clin Orthop Relat Res. 2009 Oct;467(10):2606-12. doi: 10.1007/s11999-009-0834-6. Epub 2009 Apr 10. PMID 19360453
- [Background] Learmonth ID, Young C, Rorabeck C. The operation of the century: total hip replacement. Lancet. 2007 Oct 27;370(9597):1508-19. doi: 10.1016/S0140-6736(07)60457-7. PMID 17964352
- [Background] Dieppe P, Lim K, Lohmander S. Who should have knee joint replacement surgery for osteoarthritis? Int J Rheum Dis. 2011 May;14(2):175-80. doi: 10.1111/j.1756-185X.2011.01611.x. PMID 21518317
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Hawker GA, Badley EM, Borkhoff CM, Croxford R, Davis AM, Dunn S, Gignac MA, Jaglal SB, Kreder HJ, Sale JE. Which patients are most likely to benefit from total joint arthroplasty? Arthritis Rheum. 2013 May;65(5):1243-52. doi: 10.1002/art.37901. PMID 23459843
- [Background] Wylde V, Jeffery A, Dieppe P, Gooberman-Hill R. The assessment of persistent pain after joint replacement. Osteoarthritis Cartilage. 2012 Feb;20(2):102-5. doi: 10.1016/j.joca.2011.11.011. Epub 2011 Nov 30. PMID 22178464
- [Background] Ravi B, Croxford R, Reichmann WM, Losina E, Katz JN, Hawker GA. The changing demographics of total joint arthroplasty recipients in the United States and Ontario from 2001 to 2007. Best Pract Res Clin Rheumatol. 2012 Oct;26(5):637-47. doi: 10.1016/j.berh.2012.07.014. PMID 23218428
- [Background] Ibrahim T, Bloch B, Esler CN, Abrams KR, Harper WM. Temporal trends in primary total hip and knee arthroplasty surgery: results from a UK regional joint register, 1991-2004. Ann R Coll Surg Engl. 2010 Apr;92(3):231-5. doi: 10.1308/003588410X12628812458572. Epub 2010 Mar 10. PMID 20223054
- [Background] Watanabe T, Ishizuki M, Muneta T, Banks SA. Knee kinematics in anterior cruciate ligament-substituting arthroplasty with or without the posterior cruciate ligament. J Arthroplasty. 2013 Apr;28(4):548-52. doi: 10.1016/j.arth.2012.06.030. Epub 2012 Oct 31. PMID 23122654
- [Background] Bell SW, Young P, Drury C, Smith J, Anthony I, Jones B, Blyth M, McLean A. Component rotational alignment in unexplained painful primary total knee arthroplasty. Knee. 2014 Jan;21(1):272-7. doi: 10.1016/j.knee.2012.09.011. Epub 2012 Nov 7. PMID 23140906
- [Background] Smith PN, Refshauge KM, Scarvell JM. Development of the concepts of knee kinematics. Arch Phys Med Rehabil. 2003 Dec;84(12):1895-902. doi: 10.1016/s0003-9993(03)00281-8. PMID 14669200
- [Background] Chalidis BE, Sachinis NP, Papadopoulos P, Petsatodis E, Christodoulou AG, Petsatodis G. Long-term results of posterior-cruciate-retaining Genesis I total knee arthroplasty. J Orthop Sci. 2011 Nov;16(6):726-31. doi: 10.1007/s00776-011-0152-1. Epub 2011 Sep 10. PMID 21909722
- [Background] Font-Rodriguez DE, Scuderi GR, Insall JN. Survivorship of cemented total knee arthroplasty. Clin Orthop Relat Res. 1997 Dec;(345):79-86. PMID 9418624
- [Background] Sabouret P, Lavoie F, Cloutier JM. Total knee replacement with retention of both cruciate ligaments: a 22-year follow-up study. Bone Joint J. 2013 Jul;95-B(7):917-22. doi: 10.1302/0301-620X.95B7.30904. PMID 23814243
- [Background] Price AJ, Waite JC, Svard U. Long-term clinical results of the medial Oxford unicompartmental knee arthroplasty. Clin Orthop Relat Res. 2005 Jun;(435):171-80. doi: 10.1097/00003086-200506000-00024. PMID 15930935
- [Background] Malchau H. Introducing new technology: a stepwise algorithm. Spine (Phila Pa 1976). 2000 Feb 1;25(3):285. doi: 10.1097/00007632-200002010-00004. No abstract available. PMID 10703097
- [Background] Malchau H, Bragdon CR, Muratoglu OK. The stepwise introduction of innovation into orthopedic surgery: the next level of dilemmas. J Arthroplasty. 2011 Sep;26(6):825-31. doi: 10.1016/j.arth.2010.08.007. Epub 2010 Oct 2. PMID 20888183
- [Background] Iwaki H, Pinskerova V, Freeman MA. Tibiofemoral movement 1: the shapes and relative movements of the femur and tibia in the unloaded cadaver knee. J Bone Joint Surg Br. 2000 Nov;82(8):1189-95. doi: 10.1302/0301-620x.82b8.10717. PMID 11132285
- [Background] Pinskerova V, Johal P, Nakagawa S, Sosna A, Williams A, Gedroyc W, Freeman MA. Does the femur roll-back with flexion? J Bone Joint Surg Br. 2004 Aug;86(6):925-31. doi: 10.1302/0301-620x.86b6.14589. PMID 15330038
- [Background] Pinskerova V, Samuelson KM, Stammers J, Maruthainar K, Sosna A, Freeman MA. The knee in full flexion: an anatomical study. J Bone Joint Surg Br. 2009 Jun;91(6):830-4. doi: 10.1302/0301-620X.91B6.22319. PMID 19483242
- [Background] Nakagawa S, Kadoya Y, Todo S, Kobayashi A, Sakamoto H, Freeman MA, Yamano Y. Tibiofemoral movement 3: full flexion in the living knee studied by MRI. J Bone Joint Surg Br. 2000 Nov;82(8):1199-200. doi: 10.1302/0301-620x.82b8.10718. PMID 11132287
- [Background] Freeman MA, Pinskerova V. The movement of the knee studied by magnetic resonance imaging. Clin Orthop Relat Res. 2003 May;(410):35-43. doi: 10.1097/01.blo.0000063598.67412.0d. PMID 12771815
- [Background] Freeman MA, Pinskerova V. The movement of the normal tibio-femoral joint. J Biomech. 2005 Feb;38(2):197-208. doi: 10.1016/j.jbiomech.2004.02.006. PMID 15598446
- [Background] Dahl J, Snorrason F, Nordsletten L, Rohrl SM. More than 50% reduction of wear in polyethylene liners with alumina heads compared to cobalt-chrome heads in hip replacements: a 10-year follow-up with radiostereometry in 43 hips. Acta Orthop. 2013 Aug;84(4):360-4. doi: 10.3109/17453674.2013.810516. Epub 2013 Jun 25. PMID 23795579
- [Background] Figved W, Dahl J, Snorrason F, Frihagen F, Rohrl S, Madsen JE, Nordsletten L. Radiostereometric analysis of hemiarthroplasties of the hip--a highly precise method for measurements of cartilage wear. Osteoarthritis Cartilage. 2012 Jan;20(1):36-42. doi: 10.1016/j.joca.2011.11.006. Epub 2011 Nov 15. PMID 22126919
- [Background] Pijls BG, Valstar ER, Nouta KA, Plevier JW, Fiocco M, Middeldorp S, Nelissen RG. Early migration of tibial components is associated with late revision: a systematic review and meta-analysis of 21,000 knee arthroplasties. Acta Orthop. 2012 Dec;83(6):614-24. doi: 10.3109/17453674.2012.747052. Epub 2012 Nov 9. PMID 23140091
- [Background] van Ijsseldijk EA, Lebel B, Stoel BC, Valstar ER, Gouzy S, Vielpeau C, Kaptein BL. Validation of the in vivo volumetric wear measurement for total knee prostheses in model-based RSA. J Biomech. 2013 Apr 26;46(7):1387-91. doi: 10.1016/j.jbiomech.2013.02.021. Epub 2013 Mar 26. PMID 23540721